CLINICAL TRIAL: NCT01966731
Title: REALIZING EFFECTIVENESS ACROSS CONTINENTS WITH HYDROXYUREA (REACH): A PHASE I/II PILOT STUDY OF HYDROXYUREA FOR CHILDREN WITH SICKLE CELL ANEMIA
Brief Title: Realizing Effectiveness Across Continents With Hydroxyurea (REACH)
Acronym: REACH
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-4221
Record Dates: First submitted 2013-10-04; First posted 2013-10-22 (Estimated); Results first posted 2020-11-09 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell Disease
Keywords: Africa
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Intervention Model Description: After enrollment, a two-month screening phase was used to perform baseline evaluations including nutritional and infectious assessments, along with supplements and treatments as deemed necessary by local guidelines (e.g., penicillin, pneumococcal immunization, Vitamin A and albendazole/mebendazole treatment per WHO recommendations, malaria prophylaxis, and iron/folate supplementation)
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydroxyurea (Experimental): After patient enrollment, a two-month pre-hydroxyurea evaluation phase will be used to perform baseline evaluations including nutritional and infectious assessments, and to provide supplements or treatments as deemed necessary. After the pre-hydroxyurea evaluation and supplementation phase, hydroxyurea dosing will be administered as a single daily dose, using capsules provided as a monthly supply in 200mg, 300mg, 400mg, or 500mg sizes.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — Hydroxyurea will begin at 15-20 mg/kg PO daily. Six months of treatment will be given at the fixed dose, followed by another six months with dose escalation (2.5-5.0 mg/kg increments every 8 weeks) as tolerated to 20-30 mg/kg/day or MTD. The dose escalation phase will continue through the 12-month evaluation, after which hydroxyurea will continue in maintenance phase until the common treatment termination date. The daily dose will be calculated using available capsule sizes and a goal of 15-20 (17.5 ± 2.5) mg/kg/day based on weight. After 6 months of treatment, hydroxyurea will be titrated according to myelosuppression, and will be increased to 20-30 mg/kg/day or the maximum tolerated dose (MTD). Hydroxyurea dose escalation will occur in 5.0 ± 2.5 mg/kg/day increments.
  Other Names: Hydrea; Droxia

SUMMARY:
REACH is a prospective, phase I/II open-label dose escalation trial of hydroxyurea for for pediatric patients with sickle cell anemia (SCA). The short-term goal is to obtain critical pilot data regarding the feasibility, safety, and benefit of hydroxyurea for children with SCA in multiple distinct research settings in Africa. Based on that information, the longer-term goal is to make hydroxyurea more widely available for children with SCA in Africa, particularly those identified with SCA through expanded newborn screening programs.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

1. To assess the feasibility of conducting a prospective research study using hydroxyurea therapy for SCA in sub-Saharan Africa (including adherence to monthly clinic visits and laboratory assessments, and medication compliance)
2. To monitor the safety of hydroxyurea therapy, specifically documenting hematological toxicities (cytopenias) and serious infections (bacterial and malarial)
3. To evaluate the benefits of hydroxyurea therapy, using both laboratory (e.g., fetal hemoglobin, hemoglobin, white blood cell count) and clinical parameters (e.g., pain, hospitalization, growth)
4. To explore the pharmacokinetic and genetic basis for any observed inter-patient variability in the clinical or laboratory response to hydroxyurea.
5. To evaluate the economic cost of providing hydroxyurea therapy in the REACH study sites.
6. To investigate the effects of hydroxyurea dose escalation on laboratory and clinical parameters

ELIGIBILITY:
Inclusion Criteria

1. Pediatric patients with documented sickle cell anemia (typically HbSS supported by hemoglobin electrophoresis, complete blood count, and peripheral blood smear)
2. Age range of 1.00-9.99 years, inclusive, at the time of enrollment
3. Weight at least 10.0 kg at the time of enrollment
4. Parent or guardian willing and able to provide written informed consent, with child's verbal assent as per local IRB/Ethics Board requirements
5. Willingness to comply with all study-related treatments, evaluations, and follow-up

Exclusion Criteria

1. Known medical condition making participation ill-advised, (e.g., acute or chronic infectious disease, HIV, or malignancy)
2. Acute or chronic severe malnutrition determined by impaired growth parameters as defined by WHO (weight for length/height or height for age >3 z-scores below the median WHO growth standards, as defined in Appendix I)
3. Pre-existing severe hematological toxicity (temporary exclusions)

   1. Anemia: Hb <4.0 gm/dL
   2. Anemia: Hb <6.0 gm/dL with ARC <100 x 109/L
   3. Reticulocytopenia: ARC <80 x 109/L with Hb <7.0 gm/dL
   4. Thrombocytopenia: Platelets <80 x 109/L
   5. Neutropenia: ANC <1.0 x 109/L
4. Blood transfusion within 60 days before enrollment (temporary exclusion)
5. Hydroxyurea use within 6 months before enrollment (temporary exclusion)

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 635 (Actual)
Dates: Start 2014-06; Primary Completion 2018-07-01 (Actual); Study Completion 2033-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Ware, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- Hospital Pediátrico David Bernardino, Luanda, Angola
- Centre Hospitalier Monkole, Kinshasa, Democratic Republic of the Congo
- KEMRI/Wellcome Trust Research, Kilifi, Kenya
- Ministry of Health Mbale Regional Hospital, Mbale, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Power-Hays A, McElhinney KE, Williams TN, Mochamah G, Olupot-Olupot P, Paasi G, Reid ME, Rankine-Mullings AE, Opoka RO, John CC, McGann PT, Quinn CT, Punt NC, Smart LR, Stuber SE, Latham TS, Vinks AA, Ware RE. Hydroxyurea pharmacokinetics in children with sickle cell anemia across different global populations. Blood Adv. 2026 Jan 27;10(2):418-427. doi: 10.1182/bloodadvances.2025017254. PMID 41026975
- [Derived] Aygun B, Lane A, Smart LR, Santos B, Tshilolo L, Williams TN, Olupot-Olupot P, Stuber SE, Tomlinson G, Latham T, Ware RE; REACH Investigators. Hydroxyurea dose optimisation for children with sickle cell anaemia in sub-Saharan Africa (REACH): extended follow-up of a multicentre, open-label, phase 1/2 trial. Lancet Haematol. 2024 Jun;11(6):e425-e435. doi: 10.1016/S2352-3026(24)00078-4. Epub 2024 Apr 30. PMID 38701812
- [Derived] Tshilolo L, Tomlinson G, Williams TN, Santos B, Olupot-Olupot P, Lane A, Aygun B, Stuber SE, Latham TS, McGann PT, Ware RE; REACH Investigators. Hydroxyurea for Children with Sickle Cell Anemia in Sub-Saharan Africa. N Engl J Med. 2019 Jan 10;380(2):121-131. doi: 10.1056/NEJMoa1813598. Epub 2018 Dec 1. PMID 30501550
- [Derived] McGann PT, Williams TN, Olupot-Olupot P, Tomlinson GA, Lane A, Luis Reis da Fonseca J, Kitenge R, Mochamah G, Wabwire H, Stuber S, Howard TA, McElhinney K, Aygun B, Latham T, Santos B, Tshilolo L, Ware RE; REACH Investigators. Realizing effectiveness across continents with hydroxyurea: Enrollment and baseline characteristics of the multicenter REACH study in Sub-Saharan Africa. Am J Hematol. 2018 Aug;93(4):537-545. doi: 10.1002/ajh.25034. Epub 2018 Jan 27. PMID 29318647
- [Derived] McGann PT, Tshilolo L, Santos B, Tomlinson GA, Stuber S, Latham T, Aygun B, Obaro SK, Olupot-Olupot P, Williams TN, Odame I, Ware RE; REACH Investigators. Hydroxyurea Therapy for Children With Sickle Cell Anemia in Sub-Saharan Africa: Rationale and Design of the REACH Trial. Pediatr Blood Cancer. 2016 Jan;63(1):98-104. doi: 10.1002/pbc.25705. Epub 2015 Aug 14. PMID 26275071

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydroxyurea: Hydroxyurea dosing was administered as a single daily dose, in 200mg, 300mg, 400mg, or 500mg sizes
Period: Overall Study
Arm/Group | Hydroxyurea
Started | 635
Initiated Hydroxyurea | 606
Completed 3 Months of Treatment | 600
Completed Study | 0
Completed | 0
Not Completed | 635
Not completed — Death | 2
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 2
Not completed — Follow up is not complete | 600
Not completed — Screening Failure | 29
Not completed — Found to be ineligible | 1

BASELINE CHARACTERISTICS:
Groups:
- Hydroxyurea: Hydroxyurea administered at 15-20 mg/kg/ day as a single daily dose.
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 606
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 606
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 296
  Male | 310
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 606
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 606
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Angola | 150
  Congo, The Democratic Republic of the | 156
  Uganda | 149
  Kenya | 151

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose Limiting Toxic Events
Description: An expected toxicity rate of 20% and acceptable toxicity rate of 30% were used for statistical calculations. After 53 participants at each site complete 3 months of therapy, if ≤ 15 participants have hematologic toxicity there is no early evidence against safety. If ≥ 15 of the initial participants experience toxicity, this is early evidence against safety. Future participants will begin at a lower dose of hydroxyurea (10 ± 2.5 mg/kg), with another 53 participants recruited of the same safety analysis. Upon final analysis of 133 participants at the same starting dose, safety for fixed-dose hydroxyurea can be concluded.
Time Frame: 3 months
Population: N= number of participants analyzed for toxicity during the first 3 months of trial therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 532
percentage of participants | 5.1 [3.5 to 7.3]

2. Secondary Outcome: Efficacy of Hydroxyurea
Description: The efficacy of hydroxyurea will be primarily assessed through fetal hemoglobin (HbF), comparing treatment with baseline values. Additional measures of laboratory efficacy will include changes in Hb, MCV, WBC, ANC, ARC, and bilirubin. Clinical events such as vaso-occlusive pain will be captured as secondary outcomes.
Time Frame: Assessed every 4 ± 1 weeks up to 204 months
Reporting Status: Not Posted, anticipated posting 2035-07

3. Secondary Outcome: Medication Adherence and the Ability for Families to Adhere to Monthly Clinic Visits Are Important Feasibility Outcomes
Description: Hydroxyurea treatment will be dispensed only 35 days at a time, requiring a clinic visit every 4 ± 1 weeks. Medication adherence and the ability for families to adhere to monthly clinic visits are important feasibility outcomes
Time Frame: Assessed every 4 ± 1 weeks up to 204 months
Reporting Status: Not Posted, anticipated posting 2035-07

ADVERSE EVENTS:
Time Frame: 67 months
Arm/Group | Hydroxyurea
All-Cause Mortality (participants affected / at risk) | 16/635
Serious Adverse Events (participants affected / at risk) | 66/635
Other Adverse Events (participants affected / at risk) | 500/635
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxyurea (N=635)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Splenic sequestration (Blood and lymphatic system disorders) | 8 (9)
Vaso-occlusive pain (Blood and lymphatic system disorders) | 8 (8)
Death NOS (General disorders) | 2 (2)
Fever NOS (General disorders) | 2 (2)
Bone infection (Infections and infestations) | 3 (3)
Infection unidentified (Infections and infestations) | 2 (2)
Malaria (Infections and infestations) | 12 (12)
Sepsis (Infections and infestations) | 12 (12)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Stroke (Nervous system disorders) | 10 (10)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 8 (8)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxyurea (N=635)
Vaso-occlusive pain (Blood and lymphatic system disorders) | 353 (755)
Fever NOS (General disorders) | 175 (258)
Infection unidentified (Infections and infestations) | 72 (97)
Malaria (Infections and infestations) | 216 (376)
Sepsis (Infections and infestations) | 37 (41)
Skin Infection (Infections and infestations) | 114 (184)
Upper respiratory infection (Infections and infestations) | 218 (414)
Aspartate aminotransferred (Investigations) | 37 (39)
Blood bilirubin increased (Investigations) | 44 (52)
Hemoglobin decreased (Investigations) | 239 (451)
Neutrophil count decreased (Investigations) | 41 (49)
Platelet count decreased (Investigations) | 68 (106)
Reticulocyte count decreased (Infections and infestations) | 63 (75)
Acute chest pain (Respiratory, thoracic and mediastinal disorders) | 59 (75)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT01966731/Prot_002.pdf
  • Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT01966731/SAP_003.pdf